CLINICAL TRIAL: NCT05455593
Title: Efficacy of the Combination of Water Aerobics and Metacognitive Training (MCT) on Psychological and Physical Health Variables and Their Relationship With SP1 and SP4 Biomarkers in People With Psychosis
Brief Title: Effectiveness of the Combination of Water Aerobics and Metacognitive Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Parc Sanitari Sant Joan de Déu (Other); Solidaritat Sant Joan de Déu (Unknown); Fluidra (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PIC-155-21
Record Dates: First submitted 2022-06-13; First posted 2022-07-13 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blind to the intervention recieved by the participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Water aerobics (Active Comparator): Aerobic exercises performed in a swimming pool.
  Interventions: Behavioral: Water aerobics
- Metacognitive Training (MCT) (Active Comparator): Treatment program for psychosis based on Cognitive-behavioral therapy (CBT), cognitive remediation (CRT) and psychoeducation.
  Interventions: Behavioral: Metacognitive Training (MCT)
- Combined intervention (water aerobics + MCT) (Experimental): Combination of water aerobics and MCT sessions.
  Interventions: Behavioral: Combined intervention

INTERVENTIONS:
Behavioral: Water aerobics — 1-hour session of water aerobics per week, for 3 months. A specialized trainer will carry out water aerobics sessions and will focus on motor coordination, strength and cardiovascular workout.
  Arms: Water aerobics
Behavioral: Metacognitive Training (MCT) — 1-hour session of MCT per week, for 3 months. A trained psychologist will carry out the MCT sessions. MCT addresses the most common cognitive biases in psychosis. Each session will focus on one topic, such as attributional style, jumping to conclusions, theory of mind, emotion recognition, memory or empathy.
  Arms: Metacognitive Training (MCT)
Behavioral: Combined intervention — Patients in this arm will participate in both in water aerobics and MCT sessions, once a week for each intervention.
  Arms: Combined intervention (water aerobics + MCT)

SUMMARY:
The objective of this study is to assess the efficacy of a combined intervention of water aerobics and Metacognitive Training (MCT), compared to each intervention separately, in people with psychosis. One purpose is to analyze the improvement of clinical, cognitive, metacognitive and psychosocial variables, motor coordination and physical health condition. Another purpose is to study the changes in SP1 and SP4 biomarker transcription levels as a function of the intervention received. The hypothesis is that the combined intervention will enhance the benefits of each intervention separately, specifically in symptoms, cognition, metacognition and psychosocial variables.

ELIGIBILITY:
Inclusion Criteria:

* Presence of one of the following diagnoses according to DSM-V criteria: schizophrenia, unspecific psychotic disorder, schizoaffective disorder, delusional disorder, brief psychotic disorder, schizophreniform disorder.
* Psychopatological stability
* 18 to 55 years old
* Interested in participating in both water aerobics and MCT groups

Exclusion Criteria:

* Head injury or intellectual disabillity (premorbid IQ <=70)
* Present scores on the PANSS >=5 in hostility, lack of cooperation or suspiciousness, to guarantee a good relationship in the group
* Patients with substance dependence disorder
* Problems related to water activities (phobia, severe mobility problems...)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-08-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline BCIS Beck Cognitive Insight Scale at 3 months (Beck et al., 2004; Gutierrez-Zotes et al., 2012) | Baseline and 3-month follow-up
  Cognitive insight self-registered measure (15 items): ability to analyze one's own beliefs and judgments. Self-reflectivness subscale: higher scores indicate a greater ability to reflect on one's own thoughts. Selfcertainty subscale: higher scores indicate a greater tendency to overestimate one's own beliefs without considering alternative explanations. Composite index: higher scores indicate a greater cognitive insight.
Change from Baseline Beads Task at 3 months (Brett-Jones et al., 1987) | Baseline and 3-month follow-up
  Measure of jumping to conclusions bias. It includes two tasks in which two jars with colored beads are presented. The first task has a 85:15 proportion and the second task has a 60:40 proportion. In the third task, the jars contain positive and negative comments, with a proportion of 60:40 in each jar. The person has to infer from which jar the beads or comments are drawn. Jumping to conclusions bias is present when the participant decides after seeing up to two beads or comments.
Change from Baseline CBQ Cognitive Bias Questionnaire at 3 months (Peters et al, 2013; Gutiérrez-Zotes, 2021) | Baseline and 3-month follow-up
  Measure of five cognitive biases (30 items): jumping to conclusions, intentionalising, catastrophising, emotional reasoning, and dichotomous thinking.
Change from Baseline Stress Test at 3 months | Baseline and 3-month follow-up
  Assessment of clinical and sports records, cardiorespiratory and locomotor system examination, electrocardiogram and ergometry.
Change from Baseline Molecular measures at 3 months | Baseline and 3-month follow-up
  Protein levels of SP1 and SP4 biomarkers transcription factor levels in peripheral blood mononuclear cells (PBMCs). mRNA expression levels of SP1 and SP4 biomarkers transcription factors in PBMCs.

SECONDARY OUTCOMES:
Change from Baseline PANSS Positive and Negative Syndrome Scale at 3 months (Kay et al., 1987; Peralta y Cuesta, 1995) | Baseline and 3-month follow-up
  Semi-structured interview to assess positive, negative and general symptoms of psychosis. Higher scores indicate greater severity of symptoms.
Change from Baseline BDI-II Beck Depression Inventory-II at 3 months (Beck et al., 1996) | Baseline and 3-month follow-up
  Depressive symptoms
Change from Baseline Rosenberg self-esteem scale at 3 months (Martín Albó et al, 2007) | Baseline and 3-month follow-up
  Self-esteem measure with 10 items (scores 0 to 30). Higher scores indicate greater self-esteem. Scores below 15 may indicate problematic low self-esteem.
Change from Baseline IPSAQ Internal, Personal and Situational Attributions Questionnaire at 3 months (McArthur, 1972; Bentall et al, 1991; Diez-Alegría, 2006) | Baseline and 3-month follow-up
  Attributional Style, including externalizing and personalizing bias subscales.
Change from Baseline Hinting Task at 3 months (Corcoran, Mercer & Frith, 1995) | Baseline and 3-month follow-up
  Theory of mind
Change from Baseline Faces test at 3 months (Baron Cohen, 1997; Huerta-Ramos et al., 2021) | Baseline and 3-month follow-up
  Facial emotion recognition
Change from Baseline MATRICS Consensus Cognitive Battery at 3 months (Nuechterlein et al., 2008; Rodriguez-Jimenez et al., 2012) | Baseline and 3-month follow-up
  Verbal processing speed, verbal fluency, attention, working memory, verbal learning and memory, visual learning and memory, reasoning, problem solving.
WAIS-IV (Weschler Adults Intelligence Scale, 1955) | Baseline
  Premorbid IQ assessed with the Vocabulary subscale
Change from Baseline GAF Global Assessment of Functioning at 3 months (Endicot et al., 1976) | Baseline and 3-month follow-up
  General functioning in a scale of 0-100
Change from Baseline WHO-DAS 12, Psychiatric Disability Assessment Schedule at 3 months (WHO, 1988; Vázquez-Barquero JL, 2000) | Baseline and 3-month follow-up
  Self-administered 12-item disability assessment
Change from Baseline SSQ Self Stigma Questionnaire at 3 months (Ochoa et al., 2015) | Baseline and 3-month follow-up
  Self-administered 14-item scale to assess self-stigma
Change from Baseline EuroQoL EQ-5D at 3 months (Badia et al., 1999) | Baseline and 3-month follow-up
  Self-administered 5-item to assess general quality of life
Change from Baseline SUMD Scale to Assess Unawareness of Mental Disorder at 3 months (Amador X.F., et al.; 1993; Ruiz A., et al., 2008) | Baseline and 3-month follow-up
  3 items to assess awareness of having a mental illness, awareness of medication effects and awareness of social consequences of having a mental illness, in a scale of 0-15. Higher scores mean a worse outcome.
Change from Heart Rate at 3 months | Baseline and 3-month follow-up
  Beats per minute (bpm)
Change from Blood Pressure at 3 months | Baseline and 3-month follow-up
  Millimetre of mercury (mmHg)
Change from Weight at 3 months | Baseline and 3-month follow-up
  Kilogram (Kg)
Change from Height at 3 months | Baseline and 3-month follow-up
  Centimetre (cm)
Change from Body Mass Index (BMI) at 3 months | Baseline and 3-month follow-up
  Weight and height will be combined to report BMI in kg/m^2
Change from Body Abdominal Girth at 3 months | Baseline and 3-month follow-up
  Centimetre (cm)
Change from Glucose Levels at 3 months | Baseline and 3-month follow-up
  Milligrams per decilitre (mg/dL)
Change from Total Cholesterol at 3 months | Baseline and 3-month follow-up
  Milligrams per decilitre (mg/dL)
Change from HDL Cholesterol at 3 months | Baseline and 3-month follow-up
  Milligrams per decilitre (mg/dL)
Change from LDL Cholesterol at 3 months | Baseline and 3-month follow-up
  Milligrams per decilitre (mg/dL)
Change from International Physical Activity Questionnaire (IPAQ; Booth, 2000) at 3 months | Baseline and 3-month follow-up
  Intensity of physical activity and sitting time
Change from Oviedo Sleep Questionnaire (OSQ; Bobes et al., 2000) at 3 months | Baseline and 3-month follow-up
  Sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Susana Ochoa, PhD, Principal Investigator — Parc Sanitari Sant Joan de Deu
Locations (1):
- Parc Sanitari Sant Joan de Déu, Sant Boi de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ochoa S, Verdaguer-Rodriguez M, Batlle N, Garreta F, Garcia B, Haro JM, Vila-Andreu E, Hernandez MJ, Escandell MJ, Munoz A, Vilamala S, Marcos S, Bassolas L, Pascua M, Ramos B; Thalassa Research Group. Efficacy of the combination of water aerobics and metacognitive training on psychological and physical health variables and their relationship with SP1 and SP4 biomarkers in people with psychosis: a study protocol. Front Psychol. 2024 Jun 11;15:1360004. doi: 10.3389/fpsyg.2024.1360004. eCollection 2024. PMID 38919799